CLINICAL TRIAL: NCT01626430
Title: Acute Effects of Tocotrienols on Insulinaemic and Inflammatory Responses in Metabolic Syndrome Subjects
Brief Title: Acute Effects of Tocotrienols on Insulin Sensitivity and Metabolic Risk Markers in Individuals at Risk for Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: A004/11
Record Dates: First submitted 2012-06-16; First posted 2012-06-22 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Metabolic Syndrome
Keywords: Gamma delta TRF; Insulin sensitivity; Postprandial lipaemia; Inflammatory markers; NF-κB
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 200 mg gd-TRF (Experimental)
  Interventions: Dietary Supplement: Gamma delta TRF
- 400 mg gd-TRF (Experimental)
  Interventions: Dietary Supplement: Gamma delta TRF
- Placebo (Experimental)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Gamma delta TRF — 50g of high fat meal will be given in a form of muffin and milkshake. A 200 mg, 400 mg gamma delta TRF or placebo will be incorporated into milkshake.
  Arms: 200 mg gd-TRF; 400 mg gd-TRF
Dietary Supplement: Placebo — 50g of high fat meal will be given in a form of muffin and milkshake. A 200 mg, 400 mg gamma delta TRF or placebo will be incorporated into milkshake.
  Arms: Placebo

SUMMARY:
Objectives: To compare the acute effects of gamma delta rich tocotrienol fractions (gd-TRF) on insulin sensitivity, metabolic risk markers and postprandial lipemia in individuals at risk for metabolic syndrome.

Hypothesis: Gamma delta-rich TRF will improve insulin sensitivity, metabolic risk markers and postprandial lipemia in individuals at risk for metabolic syndrome.

DETAILED DESCRIPTION:
A randomised, double-blind, crossover trial will be undertaken to test the acute effects of supplementation of 200 mg, 400 mg gd-TRF vs. placebo. There are 3 occasions for subjects to attend during postprandial period and these occasions will be separated by at least one week. On the day preceding the postprandial high fat meal challenge, subjects will be asked to avoid food high in fat, alcohol, caffeine and taking part in any strenuous exercise. Subjects will be provided with a standardised low fat meal (containing < 10 g fat) on the day preceding the postprandial study days to consume as their evening meal. They will be asked to fast overnight and instructed to avoid eating or drinking anything, except water, after 10 pm. Fasting blood samples will be collected on the next day and subjects will then consume the test meal, containing 50 g test fat supplemented with gd-TRF. Further venous blood samples will be collected at regular intervals for up to 6 hours postprandially.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-60 years
* BMI ≥ 25 kg/m2
* Elevated triacylglycerols ≥ 1.70 mmol/L
* Low HDL cholesterol < 1.04 mmol/L (men), < 1.30 mmol/L (women)
* Elevated blood pressure ≥ 130/ ≥ 85 mmHg
* Fasting plasma glucose ≥ 5.60 - 7.00 mmol/L
* Increased waist circumference ≥ 90 cm (men), ≥ 80 cm (women)

Exclusion Criteria:

* BMI ≤ 18.5 kg/m2
* Current use of antihypertensive or lipid lowering, insulin/glucose modulating medication
* Lactose/milk intolerance
* Alcohol intake exceeding a moderate intake (> 28 units per week)
* Smoker
* Pregnancy or lactation
* Fever, cold and infection during bleeding day

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
C-peptide | 0, 15, 30, 60, 90, 120, 180, 240, 300, 360 min

SECONDARY OUTCOMES:
Insulin sensitivity (insulin, glucose) | 0, 5, 15, 30, 60, 90, 120, 180, 240, 300, 360 min
Non-esterified fatty acid (NEFA) | 0, 5, 15, 30, 60, 90, 120, 180, 240, 300, 360 min
Serum triglycerides (TAG) | 0, 60, 120, 180, 240, 300, 360 min
Inflammatory markers (IL-6, IL-1β, TNF-α) | 0, 120, 240, 360 min
PBMC nuclear factor-κappa B (NF-κB) | 0, 240, 360 min

CONTACTS AND LOCATIONS:
Overall Officials: Dr Teng Kim Tiu, PhD, Principal Investigator — Malaysia Palm Oil Board
Locations (2):
- Malaysia (2):
  - Malaysia Palm Oil Board, Kajang, Selangor
  - Malaysian Palm Oil Board (MPOB), Kajang, Selangor